CLINICAL TRIAL: NCT01338025
Title: Evaluation of 3TC or FTC Mono-therapy Compared to Continuing HAART as a Bridging Antiretroviral Strategy in Persistently Non-adherent Children, Adolescents, and Young Adults Who Are Failing HAART and Have the M184V Resistance Mutation.
Brief Title: Evaluation of 3TC or FTC Mono-therapy Compared to Continuing HAART as a Bridging Strategy
Acronym: P1094
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was halted for lack of accrual
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT P1094; U01AI068632 (NIH)
Record Dates: First submitted 2011-04-16; First posted 2011-04-19 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-10

CONDITIONS: HIV Disease
Keywords: HIV; Bridging; Strategy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lamivudine; Emtricitabine; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A, non-suppressive HAART regimen (Active Comparator): In Step 1, subjects were randomized to continue their non-suppressive HAART regimen.
  In Step 2, subjects either began a new HAART regimen, continued randomized treatment, or discontinued therapy while remaining on follow-up, as decided by their provider.
  Interventions: Drug: HAART regimen
- Arm B, 3TC or FTC monotherapy (Active Comparator): In step 1, subjects were randomized to receive 3TC or FTC (the choice of 3TC or FTC was left to the provider).
  In Step 2, subjects either began a new HAART regimen, continued randomized treatment, or discontinued therapy while remaining on follow-up, as decided by their provider.
  Interventions: Drug: 3TC or FTC monotherapy

INTERVENTIONS:
Drug: HAART regimen — The study participant continued their non-suppressive HAART regimen as prescribed by their primary provider.
  Other Names: Highly active antiretrovial therapy (HAART)
  Arms: Arm A, non-suppressive HAART regimen
Drug: 3TC or FTC monotherapy — The study participant was assigned to either 3TC or FTC monotherapy (the choice of 3TC or FTC was left to the provider.
  Other Names: Lamivudine (3TC); emtricitabine (FTC)
  Arms: Arm B, 3TC or FTC monotherapy

SUMMARY:
The purpose of this study was to compare the use of lamivudine (3TC) or emtricitabine (FTC) alone vs. continuing a failing highly active antiretroviral therapy (HAART) regimen in HIV infected children, adolescents and young adults. The study was to see if there were changes in the HIV virus and if there were differences in immune function, viral load and medication side effects between the two groups over 28 weeks. Participants were assigned to either take 3TC or FTC alone or continue on his/her current failing HAART regimen. During the first 28 weeks of this study, if the participant was randomized to the continue HAART arm, he/she was not switched to a different or new, potentially suppressive HAART regimen, but continued on the current failing HAART regimen. However, if continuing HAART, the participant might be switched to a new regimen if their provider felt that it was clinically needed or the participant met certain study endpoints (e.g., drop in CD4, increase in viral load).

At the end of 28 weeks, the participant had the choice of remaining on the assigned study group medication(s) or starting a new HAART regimen prescribed by his/her doctor. Then, they would be followed for another 24 weeks to compare the difference in immune function, viral load and medication side effects between the different groups.

DETAILED DESCRIPTION:
Currently, there is no clear consensus for managing virologic failure. Generally, failure of non-nucleoside reverse transcriptase inhibitor (NNRTI)-based therapy due to non-adherence is associated with high rates of NNRTI resistance, while failure of protease inhibitor (PI)-based therapy due to non-adherence carries a much lower risk of PI resistance. In the setting of incomplete adherence and virologic failure despite adherence education, an optimal strategy would be one that effectively bridges the period between the cessation of the failing regimen of highly active antiretroviral (ARV) therapy and initiation of a new HAART regimen. This would provide time for interventions to improve adherence to be effective while minimizing accumulation of additional drug resistance mutations. Given the compelling need for an effective bridging strategy, the limited evidence for the safety and efficacy of this bridging regimen, and the high level of acceptability of studying 3TC or FTC monotherapy as an effective alternative, P1094 proposed to conduct a randomized clinical trial (RCT) comparing use of 3TC or FTC monotherapy as a short-term bridging regimen vs. continuation of non-suppressive HAART in non-adherent subjects.

This study closed early due to lack of accrual, with only 33 of the target 344 participants enrolled. Therefore analyses, including the analysis of the primary outcome, are descriptive. Only analyses for Step 1 could be done (Step 2 was observational). The following secondary analyses could not be performed:

Changes in Genotypic HIV Drug Resistance From Baseline Changes HIV Replication Capacity [Time Frame: 28 and 52 weeks] Changes in CD4 Percent and CD4+ T Cell Count [Time Frame: 52 weeks] Changes in HIV-1 RNA Levels [Time Frame: 52 Weeks] Changes in Immune Activation [Time Frame: 28 and 52 Weeks] Number and Percent of Subjects With Adverse Clinical Outcomes [Time Frame: 52 Weeks] Adherence as Measured by 3-day Recall [Time Frame: 52 Weeks]

ELIGIBILITY:
Step 1 Inclusion Criteria:

* Age greater than or equal to 8 to less than 25 years of age, at study entry
* Documentation of HIV-1 infection defined as positive results from two samples collected at different time points
* Treatment experienced patients must have demonstrated failure on the current HAART regimen for 2 months or longer. These patients must have been on ARVs for at least a total of 6 months prior to entry. Thus, if the failing regimen was the first ARV regimen, then the patient must have been on that initial regimen for a minimum of 6 months total.
* CD4+ T cell count greater than or equal to 100 cells/mm3 (confirmed on at least two occasions within 6 months of study entry, including the screening value)
* Documentation of the M184V mutation on genotypic testing at any time prior to study entry
* In the best judgment of the clinical site team, concerns about the subject's ability to adhere made it unsuitable to initiate a new optimal HAART regimen for at least 6 months.
* Subject had not become adherent despite site's adherence interventions
* Female subjects of reproductive potential engaging in sexual activity that could lead to pregnancy had to agree to avoid pregnancy during the entire 52 week trial and to consistently and appropriately use at least two of the following contraception methods: condoms, diaphragm or cervical cap with spermicide, IUD, hormonal-based contraception. A list of acceptable methods can be found at the FDA Birth Control Guide (http://www.fda.gov/womens).
* Parent/legal guardian or subject able and willing to provide signed informed consent when applicable

Step 1 Exclusion Criteria:

* Positive hepatitis B surface antigen or known active hepatitis B infection.
* Pregnant or breastfeeding.
* Active malignancy within the past 2 years.
* Current immunosuppressive therapy, including the equivalent of greater than 1 mg/kg/per day or greater than 20 mg total daily dose of prednisone in the 2 weeks preceding screening. Subjects for whom long-term systemic corticosteroid therapy (greater than 2 weeks) was anticipated were excluded. [Note: non-steroidal anti-inflammatory agents and inhaled, nasal, and topical corticosteroids were not excluded as immunosuppressive therapy.]
* Prior immunization with an HIV-specific vaccine
* Greater than or equal to 1 CDC class C event within the past 12 months.
* Renal disease (as defined by estimated creatinine clearance less than 50 mL/min/1.73m2 confirmed on two occasions within 3 months of screening).
* Active opportunistic infections, including active tuberculosis (TB).
* Current treatment for active systemic TB. If recent, infection must have completed treatment course. INH treatment for latent TB is allowed.
* Viral load greater than 250,000 copies/mL at screening.
* Known greater than or equal than Grade 3 of any of the following laboratory toxicities within 30 days prior to study entry: neutrophil count, hemoglobin, platelets, AST, ALT, lipase, serum creatinine. Note: Subjects could be re-screened and enrolled if repeat value was less than Grade 3 without signs or symptoms of related organ dysfunction.
* Known greater than or equal to Grade 4 laboratory toxicities within 30 days prior to study entry, except with approval of the study team.
* For subjects who were not taking 3TC or FTC at the time of screening: Documented prior intolerance or adverse effect reasonably attributed to 3TC or FTC that resulted in permanent discontinuation.
* Problems with non-adherence attributed to modifiable structural barriers, such as lack of resources (e.g., insurance, transportation).

Step 2 - Inclusion Criteria

* Met requirements for completion of Step 1
* Subject/guardian agree to continue participation in Step 2
* ViroSeq assay results had been received by site and reviewed by investigator

Ages: 8 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison L. Agwu, MD, Sc.M., Study Chair — Johns Hopkins University
Locations (17):
- United States (10):
  - Univ. of California San Francisco NICHD CRS (5091), San Francisco, California
  - Children's National Med. Ctr. Washington DC NICHD CRS (5015), Washington D.C., District of Columbia
  - University of Florida (5051), Jacksonville, Florida
  - Univ of Miami Pediatric/Perinatal HIV/AIDS (4201), Miami, Florida
  - Chicago Children's CRS (4001), Chicago, Illinois
  - Johns Hopkins University NICHD CRS (5092), Baltimore, Maryland
  - Metropolitan Hospital (5003), New York, New York
  - SUNY Stony Brook NICHD CRS (5040), Stony Brook, New York
  - Bronx-Lebanon Hospital (6901), The Bronx, New York
  - DUMC Ped. CRS (4701), Durham, North Carolina
- Hospital General de Agudos Buenos Aires Argentina NICHD CRS (5082), Buenos Aires, Argentina
- Brazil (3):
  - Hospital Geral De Nova Igaucu Brazil NICHD CRS (5097), Rio de Janeiro, Rio de Janeiro
  - Insituto de Infectologia Emilio Ribas NICHD CRS (5075), São Paulo
  - Univ of Sao Paulo Brazil NICHD CRS (5074), São Paulo
- University of Puerto Rico Pediatric HIV/AIDS Research (6601), San Juan, Puerto Rico
- Thailand (2):
  - Siriraj Hospital Mahidol University CRS (8251), Bangkok, Ratchathewi,
  - Chiang Mai University Pediatrics-Obstetrics CRS (20101), Chiang Mai

REFERENCES:
- [Derived] Agwu AL, Warshaw MG, McFarland EJ, Siberry GK, Melvin AJ, Wiznia AA, Fairlie L, Boyd S, Harding P, Spiegel HML, Abrams EJ, Carey VJ; P1094 Study Team. Decline in CD4 T lymphocytes with monotherapy bridging strategy for non-adherent adolescents living with HIV infection: Results of the IMPAACT P1094 randomized trial. PLoS One. 2017 Jun 12;12(6):e0178075. doi: 10.1371/journal.pone.0178075. eCollection 2017. PMID 28604824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 17 sites in the United States, Argentina, Brazil and Thailand. Enrollment occurred from May 10, 2011 to January 16, 2013.
Pre-assignment Details: Eligible participants were HIV-infected, ≥8 to <25 years of age with documentation of the M184V HIV resistance mutation, were failing their current antiretroviral regimen and were persistently non-adherent. Participants were randomized equally to the two study arms.
Groups:
- Arm A, Non-suppressive HAART Regimen: In Step 1, subjects were randomized to continue their non-suppressive HAART regimen.
  In Step 2, subjects either began a new HAART regimen, continue randomized treatment, or discontinued therapy while remaining on follow-up, as decided by their provider.
  HAART regimen: The study participant continued their non-suppressive HAART regimen as prescribed by their primary provider.
- Arm B, 3TC or FTC Monotherapy: In step 1, subjects were randomized to receive 3TC or FTC (the choice of 3TC or FTC was left to the provider.) In Step 2, subjects either began a new HAART regimen, continue randomized treatment, or discontinue therapy while remaining on follow-up, as decided by their provider.
  3TC or FTC monotherapy: The study participant was assigned to either 3TC or FTC monotherapy (the choice of 3TC or FTC was left to the provider.)
Period: Overall Study
Arm/Group | Arm A, Non-suppressive HAART Regimen | Arm B, 3TC or FTC Monotherapy
Started | 16 | 17
Completed | 5 | 6
Not Completed | 11 | 11
Not completed — Unexpected closure of study | 10 | 9
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Found ineligible after starting | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants who entered the study were included in analyses. One participant on Arm A did not meet entry eligibility criteria; was taken off study after the entry visit, and is therefore excluded from all analyses.
Groups:
- Arm A, Non-suppressive HAART Regimen: In Step 1, subjects will be randomized to continue their non-suppressive HAART regimen as prescribed by their primary provider.
  In Step 2, subjects will either begin a new HAART regimen, continue randomized treatment, or discontinue therapy while remaining on follow-up, as decided by their provider.
- Arm B, 3TC or FTC Monotherapy: In step 1, subjects will be randomized to receive 3TC or FTC (the choice of 3TC or FTC will be left to the provider).
  In Step 2, subjects will either begin a new HAART regimen, continue randomized treatment, or discontinue therapy while remaining on follow-up, as decided by their provider.
- Total: Total of all reporting groups
Arm/Group | Arm A, Non-suppressive HAART Regimen | Arm B, 3TC or FTC Monotherapy | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 11 | 18
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
  Argentina | 2 | 1 | 3
  Brazil | 1 | 4 | 5
  Thailand | 3 | 3 | 6
Screening CD4 count [Mean (Standard Deviation); unit: cells/mm3] | 509 (176) | 511 (277) | 510 (232)
HIV-1 RNA viral load [Mean (Standard Deviation); unit: log10 copies/mL] | 4.0 (1.0) | 3.8 (0.7) | 3.9 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immunologic Deterioration
Description: Immunologic deterioration was declared for a participant if any one of the following conditions is observed within the first 28 weeks:
  * greater than or equal to 30% decline in absolute CD4+ T cell count from entry, or
  * development of CDC class C events.
  Results report number of participants with immunologic deterioration at week 28 calculated.
Time Frame: From entry to week 28
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Arm A, Non-suppressive HAART Regimen: In Step 1, subjects will be randomized to continue their non-suppressive HAART regimen.
  In Step 2, subjects will either begin a new HAART regimen, continue randomized treatment, or discontinue therapy while remaining on follow-up, as decided by their provider.
  HAART regimen: The study participant will continue their non-suppressive HAART regimen as prescribed by their primary provider.
- Arm B, 3TC or FTC Monotherapy: In step 1, subjects will be randomized to receive 3TC or FTC (the choice of 3TC or FTC will be left to the provider).
  In Step 2, subjects will either begin a new HAART regimen, continue randomized treatment, or discontinue therapy while remaining on follow-up, as decided by their provider.
  3TC or FTC monotherapy: The study participant will be assigned to either 3TC/FTC monotherapy (the choice of 3TC or FTC will be left to the provider.
Arm/Group | Arm A, Non-suppressive HAART Regimen | Arm B, 3TC or FTC Monotherapy
Number analyzed (Participants) | 15 | 17
participants | 0 | 5
Statistical Analysis 1: Comparison: Arm A, Non-suppressive HAART Regimen vs Arm B, 3TC or FTC Monotherapy; Test type: Superiority or Other; p = 0.03, Log Rank

2. Secondary Outcome: Change in CD4+ T Cell Count
Description: Change in CD4+ T cell count from entry to Week 28 (CD4+ at entry - CD4+ at Week 28).
Time Frame: Entry to week 28
Population: All eligible participants with CD4+ cell count results available at entry and at week 28.
Measure: Median (Inter-Quartile Range); unit: CD4+ T cell count/mL
Arm/Group | Arm A, Non-suppressive HAART Regimen | Arm B, 3TC or FTC Monotherapy
Number analyzed (Participants) | 6 | 8
CD4+ T cell count/mL | 27.5 [-44 to 45] | 76 [1.5 to 222]

3. Secondary Outcome: Change in HIV-1 RNA Levels
Description: Change in HIV-1 RNA levels from Entry to Week 28
Time Frame: 28 Weeks
Population: All eligible participants with HIV-1 RNA results available at entry and at week 28.
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Arm A, Non-suppressive HAART Regimen | Arm B, 3TC or FTC Monotherapy
Number analyzed (Participants) | 8 | 6
copies/mL | 3087 [-3,000 to 17,761] | -2241 [-20,354 to -680]

4. Secondary Outcome: Number of Participants Non-adherent as Measured by 3-day Recall
Description: Number of participants reporting a missed medication dose in the past 3 days.
Time Frame: 28 Weeks
Population: All eligible participants with adherence data available at week 28.
Measure: Number; unit: participants
Arm/Group | Arm A, Non-suppressive HAART Regimen | Arm B, 3TC or FTC Monotherapy
Number analyzed (Participants) | 6 | 7
participants | 3 | 1

ADVERSE EVENTS:
Time Frame: From study enrollment until study completion or discontinuation.
Description: Expedited adverse event (AE) reporting followed requirements, definitions and methods for expedited reporting of Adverse Events (AEs) as outlined in Version 2.0 of the DAIDS EAE Manual, available on the RSC website at http://rsc.tech-res.com/safetyandpharmacovigilance/.
Arm/Group | Arm A, Non-suppressive HAART Regimen | Arm B, 3TC or FTC Monotherapy
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 15/16 | 15/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A, Non-suppressive HAART Regimen (N=16) | Arm B, 3TC or FTC Monotherapy (N=17)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Axillary pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Acarodermatitis (Infections and infestations) | 0 | 1
Body tinea (Infections and infestations) | 0 | 1
Cutaneous larva migrans (Infections and infestations) | 1 | 0
Ear infection bacterial (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Infection protozoal (Infections and infestations) | 0 | 1
Lice infestation (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Purulent discharge (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 2
Vaginitis bacterial (Infections and infestations) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase abnormal (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3
Blood alkaline phosphatase abnormal (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood bicarbonate decreased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 3 | 0
Blood cholesterol increased (Investigations) | 4 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose abnormal (Investigations) | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 0 | 2
Haemoglobin decreased (Investigations) | 1 | 1
Lipase abnormal (Investigations) | 1 | 2
Low density lipoprotein increased (Investigations) | 3 | 2
Neutrophil count decreased (Investigations) | 4 | 1
Platelet count decreased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Oppositional defiant disorder (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No